CLINICAL TRIAL: NCT05997355
Title: "Preoperative Gabapentin and Its Effects on Postoperative Analgesia in Patients Undergoing Cosmetic Breast Surgery"
Brief Title: Preoperative Gabapentin for Cosmetic Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Miguel Serpa Irizarry, MD, University of Puerto Rico
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3650222
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Treatment with gabapentin vs no treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patient will be treated with preoperative gabapentin
  Interventions: Drug: Gabapentin 600Mg Tab
- No treatment (No Intervention): Patient will not be treated with preoperative gabapentin

INTERVENTIONS:
Drug: Gabapentin 600Mg Tab — A single preoperative dose of gabapentin 600mg
  Arms: Treatment

SUMMARY:
The goal of this clinical trial is to compare postoperative pain and opioid consumption in patients who undergo cosmetic breast surgery and are treated preoperatively with gabapentin. The main questions to answer are the amount of postoperative pain on a scale of 0-10 and amount of opioids consumed postoperatively. Participants will be randomized into two groups: treatment vs no treatment. Treatment group will receive 600mg of gabapentin preopreatively. Researchers will compare treatment vs no treatment group to determine the effects of preoperative gabapentin on postoperative pain management and opioid consumption.

DETAILED DESCRIPTION:
HYPOTHESIS We hypothesize that a single dose of preoperative gabapentin will improve postoperative pain scores and decrease postoperative opioid requirements in our study population. This will be tested by administering a preoperative dose of 600mg of gabapentin and measuring pain scores and amount of opioid consumption during the postoperative period. The study will compare two groups. Participants will be randomly assigned to one of the two groups and will consist of a treatment group and a control group. We will measure pain scores in a simple 0-10 scale and amount of opioid consumption during the first 7 days after discharge and compare them with patients who did not receive preoperative gabapentin. Our aims are to determine if gabapentin improves postoperative analgesia and reduces postoperative opioid requirements in a population undergoing cosmetic breast surgery

METHODOLOGY AND STUDY DESIGN

This study will be a randomized control trial. Participants will be randomized and divided into treatment versus no treatment group. Treatment group will be administered a dose of 600mg of gabapentin within 2 hours of surgery. Amount of postoperative opioids will be measured for 7 days, post op pain scores will be measured twice daily for 7 days. This information will be collected via postoperative questionnaires.

STUDY SUBJECTS Participants will be adult, non pregnant patients older than 18 years undergoing cosmetic breast surgery at either Hospital Oncologico Isaac Gonzalez Martinez or Hospital UPR Federico Trilla. Participants will be selected during the initial clinic visit, there will be no specific recruiting strategies. Excluded populations include minors 18 years old or less as well as pregnant females due to health concerns. Participants will be explained in detail the goal and objectives of study along with risks vs benefits. The following HIPAA identifiers will be excluded: Geographical elements, fax numbers, social security numbers, health insurance beneficiary numbers, vehicle identifiers, digital identifiers, digital attributes, IP addresses, biometric elements and full face photographic images.

VARIABLES

Primary outcomes will be the amount of postoperative pain and amount of postoperative opioid consumption. Postoperative pain will be defined and measured as a score from 1-10. Opioid consumption will be defined and measured as the amount of standard doses used in the postoperative period. Prior chronic gabapentin or opioid use will also be a variable accounted for to eliminate confounding effects of tachyphylaxis.

ANALYTIC PLAN Data will be organized in tables and analyzed with simple t-test to compare mean pain scores and amount of postoperative opioid consumption. Data will be stored within a shared google drive folder in a private excel/google sheets document. Each researcher listed in the study protocol will have access to the data individually via their own electronic devices in order to access when needed. CO-PI will administer privacy settings and provide access to each researcher. Data checks will periodically be performed to ensure data consistency.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 to 65 y/o without chronic gabapentin and/or opioid use

Exclusion Criteria:

* minors less than 18 y/o, adults older than 65 y/o, chronic users of gabapentin and/or opioids, pregnant females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Days 1-7 postoperatively
  Amount of postoperative pain on a scale from 1-10
Postoperative opioid consumption | Days 1-7 postoperatively
  Amount of postoperative standardized opioid doses

CONTACTS AND LOCATIONS:
Overall Officials: Angel Rivera Barrios, MD, Principal Investigator — angel.rivera56@upr.edu

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers via a private shared online folder.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the complete duration of the study
Access Criteria: Researchers will be invited by PI or CO-PI to shared folder. Information will not be shared outside of research group nor made public

REFERENCES:
- [Background] Chang CY, Challa CK, Shah J, Eloy JD. Gabapentin in acute postoperative pain management. Biomed Res Int. 2014;2014:631756. doi: 10.1155/2014/631756. Epub 2014 Apr 14. PMID 24829909
- [Background] Seib RK, Paul JE. Preoperative gabapentin for postoperative analgesia: a meta-analysis. Can J Anaesth. 2006 May;53(5):461-9. doi: 10.1007/BF03022618. PMID 16636030
- [Background] Liu B, Liu R, Wang L. A meta-analysis of the preoperative use of gabapentinoids for the treatment of acute postoperative pain following spinal surgery. Medicine (Baltimore). 2017 Sep;96(37):e8031. doi: 10.1097/MD.0000000000008031. PMID 28906391
- [Background] Mao Y, Wu L, Ding W. The efficacy of preoperative administration of gabapentin/pregabalin in improving pain after total hip arthroplasty: a meta-analysis. BMC Musculoskelet Disord. 2016 Aug 30;17(1):373. doi: 10.1186/s12891-016-1231-4. PMID 27577678
- [Background] Hu J, Huang D, Li M, Wu C, Zhang J. Effects of a single dose of preoperative pregabalin and gabapentin for acute postoperative pain: a network meta-analysis of randomized controlled trials. J Pain Res. 2018 Nov 2;11:2633-2643. doi: 10.2147/JPR.S170810. eCollection 2018. PMID 30519075
- [Background] Rai AS, Khan JS, Dhaliwal J, Busse JW, Choi S, Devereaux PJ, Clarke H. Preoperative pregabalin or gabapentin for acute and chronic postoperative pain among patients undergoing breast cancer surgery: A systematic review and meta-analysis of randomized controlled trials. J Plast Reconstr Aesthet Surg. 2017 Oct;70(10):1317-1328. doi: 10.1016/j.bjps.2017.05.054. Epub 2017 Jun 9. PMID 28751024
- [Background] Dirks J, Fredensborg BB, Christensen D, Fomsgaard JS, Flyger H, Dahl JB. A randomized study of the effects of single-dose gabapentin versus placebo on postoperative pain and morphine consumption after mastectomy. Anesthesiology. 2002 Sep;97(3):560-4. doi: 10.1097/00000542-200209000-00007. PMID 12218520
- [Background] Freedman BM, O'Hara E. Pregabalin has opioid-sparing effects following augmentation mammaplasty. Aesthet Surg J. 2008 Jul-Aug;28(4):421-4. doi: 10.1016/j.asj.2008.04.004. PMID 19083556
- [Background] Barker JC, DiBartola K, Wee C, Andonian N, Abdel-Rasoul M, Lowery D, Janis JE. Preoperative Multimodal Analgesia Decreases Postanesthesia Care Unit Narcotic Use and Pain Scores in Outpatient Breast Surgery. Plast Reconstr Surg. 2018 Oct;142(4):443e-450e. doi: 10.1097/PRS.0000000000004804. PMID 29979365